CLINICAL TRIAL: NCT03861429
Title: Me & My Wishes: An Efficacy Trial of Long Term Care Residents With Alzheimer's Using Videos to Communicate Care Preferences With Caregivers
Brief Title: Me & My Wishes: An Efficacy Trial Using Videos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Brown University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gail Towsley, Associate Professor, University of Utah
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00111417; 1R21AG058094 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-03-04 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Health Communication

STUDY DESIGN:
Intervention Model Description: The investigators propose Stage II efficacy testing of Me & My Wishes using a randomized wait-list control design that allows the investigators to compare the effects between an early intervention group (Group 1) and a wait-list "control" group (Group 2).Six NHs matched on number of beds and payor mix will be randomly assigned to one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Me & My Wishes Intervention/Group 1 (Experimental): In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline.
  Interventions: Behavioral: Me & My Wishes
- Me & My Wishes Wait-list control/Group 2 (Other): In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be produced and viewed within three months.
  Interventions: Behavioral: Me & My Wishes

INTERVENTIONS:
Behavioral: Me & My Wishes — Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.

SUMMARY:
The aim of this study is to determine whether the Me & My Wishes intervention positively impacts communication of preferences among nursing home residents with dementia and their family caregivers and care team.

DETAILED DESCRIPTION:
Me & My Wishes are videos of nursing home residents talking about their preferences for care, including four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Knowing what residents want is essential to staff's ability to provide quality care and can inform family caregivers decision making especially in later stages of life as the resident's cognition declines-a time when family caregivers often feel unprepared. Persons with mild to moderate dementia can accurately express their everyday and EOL preferences, however, stereotypes persist about the decision making abilities of people with dementia that often prevent their involvement in conversations about care. The investigators propose to conduct a Stage II efficacy trial of Me & My Wishes-a novel approach for communicating resident care preferences-by creating videos with 48-54 nursing home residents with mild to moderate dementia and sharing their personalized video with informal (family) and formal (staff) caregivers. The investigators will employ a randomized wait-list control design in which residents in control nursing homes will delay sharing their video. Videos may be viewed two ways: 1) in resident quarterly care conferences; and 2) via a web-based link with resident-identified family members or friends.

ELIGIBILITY:
Resident Inclusion Criteria:

* Identified as having Alzheimer's or related dementia
* Mild to moderate cognitive impairment (BIMS = 8-15, (MDS C0500) (nursing home residents only)
* Makes Self Understood = <1 (MDS B0700)/present in medical record
* Understood By Others = <1 (MDS B0800)/present in medical record
* Reside at the facility at least 2 weeks identified as a long-term resident
* Age >65 years
* Speaks English

Family Inclusion Criteria:

* Speaks English
* Willing and able to watch the videos
* Willing to complete short surveys. Being unable to attend care conference to view the video (e.g. due to distance) will not exclude family from participating.

Staff Inclusion Criteria:

* Speaks English
* Willing to watch the videos
* Willing to complete short surveys

Resident Exclusion Criteria:

* Limited communication capacity (e.g. aphasia)
* Comatose
* Cognitively intact
* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Marquis Hope Village Assisted Living, Canby, Oregon
  - Marquis Forest Grove Assisted Living, Forest Grove, Oregon
  - Marquis Forest Grove Post Acute Rehab, Forest Grove, Oregon
  - Regency Gresham Nursing and Rehabilitation Center, Gresham, Oregon
  - Marquis Wilsonville Assisted Living, Wilsonville, Oregon
  - Marquis Wilsonville Post Acute Rehab, Wilsonville, Oregon
  - French Prairie Nursing and Rehab, Woodburn, Oregon
  - Woodland Care Center, Woodland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Towsley GL, Neller S, Baier RR, Wong B. Me & My Wishes: Concordance of End-of-Life Preferences between Residents with Dementia, Family, and Staff. J Palliat Med. 2022 Jun;25(6):880-887. doi: 10.1089/jpm.2021.0111. Epub 2021 Dec 28. PMID 34962157

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nursing homes, assisted living
Groups:
- Me & My Wishes Intervention/Group 1: In Group 1 (early intervention group) NHs, families, and staff video recording, editing, and viewing will occur within three months of baseline.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
- Me & My Wishes Wait-list Control/Group 2: In Group 2 (delayed sharing) NHs, residents, families, and staff will be on a wait-list; after the delayed start, their video will be produced and viewed within three months.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
Period: Overall Study
Arm/Group | Me & My Wishes Intervention/Group 1 | Me & My Wishes Wait-list Control/Group 2
Started | 64; 4 nursing homes, assisted living | 74; 4 nursing homes, assisted living
Residents | 17; 4 nursing homes, assisted living | 19; 4 nursing homes, assisted living
Family | 25; 4 nursing homes, assisted living | 25; 4 nursing homes, assisted living
Staff | 13; 4 nursing homes, assisted living | 25; 4 nursing homes, assisted living
Completed | 55; 4 nursing homes, assisted living | 69; 4 nursing homes, assisted living
Not Completed | 9; 0 nursing homes, assisted living | 5; 0 nursing homes, assisted living

BASELINE CHARACTERISTICS:
Population: Residents, family, and staff who completed the study.
Groups:
- Me & My Wishes Intervention/Group 1 Residents: In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
- Me & My Wishes Wait-list Control/Group 2 Residents: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be produced and viewed within three months.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
- Me & My Wishes Intervention/Group 1 Family: In Group 1 (early intervention group) NHs, resident's video will be shared within three months of baseline.
  Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Videos are then shared.
- Me & My Wishes Wait-list Control/Group 2 Family: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be shared with family within three months.
  Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Videos are then shared.
- Me & My Wishes Intervention/Group 1 Staff: In Group 1 (early intervention group) NHs, resident's video will be shared with staff within three months of baseline.
  Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Videos are then shared.
- Me & My Wishes Wait-list Control/Group 2 Staff: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be shared with staff within three months.
  Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Videos are then shared.
- Total: Total of all reporting groups
Arm/Group | Me & My Wishes Intervention/Group 1 Residents | Me & My Wishes Wait-list Control/Group 2 Residents | Me & My Wishes Intervention/Group 1 Family | Me & My Wishes Wait-list Control/Group 2 Family | Me & My Wishes Intervention/Group 1 Staff | Me & My Wishes Wait-list Control/Group 2 Staff | Total
Number analyzed (Participants) | 17 | 19 | 25 | 25 | 13 | 25 | 124
Age, Categorical [Count of Participants; unit: Participants] — Population: Age not reported for two participants (e.g., left blank)
  Participants
    number analyzed (Participants) | 17 | 19 | 25 | 25 | 12 | 24 | 122
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 17 | 13 | 12 | 21 | 63
    >=65 years | 17 | 19 | 8 | 12 | 0 | 3 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.77 (17.31) | 57.75 (18.24) | 59.84 (10.15) | 61.56 (12.88) | 47.33 (10.97) | 41.58 (16.83) | 60.86 (18.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 15 | 21 | 12 | 20 | 90
  Male | 8 | 6 | 10 | 4 | 1 | 5 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 1 | 5
  Not Hispanic or Latino | 16 | 17 | 24 | 24 | 13 | 23 | 117
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 0 | 1 | 0 | 1 | 6
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 2
  White | 14 | 18 | 25 | 24 | 13 | 19 | 113
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 19 | 25 | 25 | 13 | 25 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Documented Discussion of Goals of Care
Description: At each specified time point, a chart review was conducted to obtain whether goals of care discussions occurred (change in documentation in medical record, e.g. social work note), yes/no. Reported values indicated residents who had a documented GOC in chart (yes) at any time point.
  Goal of Care Conversations encompass two parts. A) some sharing of disease status / prognosis + B) discussion of a choice of goals/treatment decisions.
  Examples of Part A include disease understanding, disease state, disease progression, prognosis/life expectancy, documentation that the clinician tried to discuss prognosis but the patient/family refused
Time Frame: Baseline, time of sharing (3 months from baseline), and 90 days post sharing video
Population: persons living with dementia (PLWD) in long-term care (LTC) settings, such as nursing homes and assisted living communities
Measure: Count of Participants; unit: Participants
Groups:
- Me & My WishesIntervention/Group 1 Resident: In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
- Me & My Wishes Wait-list Control/Group 2 Resident: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be produced and viewed within three months.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
Arm/Group | Me & My WishesIntervention/Group 1 Resident | Me & My Wishes Wait-list Control/Group 2 Resident
Number analyzed (Participants) | 17 | 19
Participants | 12 | 10
Statistical Analysis 1: Comparison: Me & My WishesIntervention/Group 1 Resident vs Me & My Wishes Wait-list Control/Group 2 Resident; Multilevel logistic regression (generalized estimating equations [GEE] with an autoregressive (1) working correlation matrix, logit link function) were fitted to assess the primary hypotheses. The models account for the repeated measures (3 or 4 time points), correlated, data structure per person. An additive model was conducted with contrast coding for each time point, treatment, and follow-up effects; Test type: Superiority; p = .105, Mixed Models Analysis; Odds Ratio (OR) = 3.32, 95% CI 2-sided [.78 to 14.15]

2. Secondary Outcome: Self-efficacy for Communicating Preferences
Description: Confidence in expressing or communicating about resident preferences. Self-efficacy items, range 1-5, higher is more confident.
Time Frame: Baseline, time of sharing (3 months from baseline), and 90 days post sharing video
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Me & My Wishes Intervention/Group 1 Resident: In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline.
  Me & My Wishes: Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
Arm/Group | Me & My Wishes Intervention/Group 1 Resident | Me & My Wishes Wait-list Control/Group 2 Resident
Number analyzed (Participants) | 17 | 19
score on a scale
  Baseline | 4.26 (.13) | 4.26 (.13)
  Time of sharing | 4.37 (.15) | 3.77 (.26)
  90 day | 4.38 (.16) | 3.96 (.25)
Statistical Analysis 1: Comparison: Me & My Wishes Intervention/Group 1 Resident vs Me & My Wishes Wait-list Control/Group 2 Resident; Test type: Superiority; p = .04, Mixed Models Analysis; Mean Difference (Final Values) = .6, 95% CI 2-sided [.022 to 1.178] — Calculation of mean differences were derived from mixed model analyses

3. Other Pre Specified Outcome: Concordance of Psychosocial Preferences Between Video and Staff
Description: Psychosocial preferences include having family at the bedside; engaging in faith practices, such as prayer; having a pet at bedside; and engaging in activities such as being read to or listening to music. Preferences from the videos and surveys were coded as yes, no, don't know, or missing. Concordance occurred when the coded preferences in the resident's video and staff member response matched.
Time Frame: Baseline, time of sharing (within 3 months of baseline), and 90 days post sharing video
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Me & My Wishes Intervention/Group 1 | Me & My Wishes Wait-list Control/Group 2
Number analyzed (Participants) | 17 | 19
percentage of agreement
  Baseline | 47.87 (29.87) | 44.87 (31.82)
  Time of Sharing | 77.50 (19.45) | 87.25 (18.28)
  90 days | 68.60 (24.45) | 60.29 (30.49)
Statistical Analysis 1: Comparison: Me & My Wishes Intervention/Group 1 vs Me & My Wishes Wait-list Control/Group 2; Test type: Superiority; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = .29, 95% CI 2-sided [.12 to .46] — Calculation of mean differences were derived from mixed model analyses

4. Other Pre Specified Outcome: Concordance of End of Life Preferences, Video and Staff
Description: EOL preferences include treatment preferences (cardiopulmonary resuscitation, or CPR; breathing machine; tube feeding; life support; and pain treatment). Preferences from the videos and surveys were coded as yes, no, don't know, or missing. Concordance occurred when the coded preferences in the resident's video and staff member response matched.
Time Frame: Baseline, time of sharing (within 3 months of baseline), and 90 days post sharing video
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Me & My Wishes Intervention/Group 1 | Me & My Wishes Wait-list Control/Group 2
Number analyzed (Participants) | 17 | 19
percentage of agreement
  Baseline | 29.79 (24.98) | 27.18 (25.37)
  Time of Sharing | 63.50 (22.59) | 55.29 (28.17)
  90 days | 60.93 (23.07) | 46.27 (28.70)
Statistical Analysis 1: Comparison: Me & My Wishes Intervention/Group 1 vs Me & My Wishes Wait-list Control/Group 2; Test type: Superiority; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = .35, 95% CI 2-sided [.21 to .48] — Calculation of mean differences were derived from mixed model analyses

5. Other Pre Specified Outcome: Concordance of Psychosocial Preferences, Video and Family
Description: Psychosocial preferences include having family at the bedside; engaging in faith practices, such as prayer; having a pet at bedside; and engaging in activities such as being read to or listening to music. Preferences from the videos and surveys were coded as yes, no, don't know, or missing. Concordance occurred when the coded preferences in the resident's video and family member response matched.
Time Frame: Baseline, time of sharing (within 3 months of baseline), and 90 days post sharing video
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Me & My Wishes Intervention/Group 1 | Me & My Wishes Wait-list Control/Group 2
Number analyzed (Participants) | 17 | 19
percentage of agreement
  Baseline | 67.31 (24.26) | 64.13 (30.92)
  Time of Sharing | 72.00 (22.03) | 83.70 (23.37)
  90 days | 71.74 (24.20) | 85.53 (19.21)
Statistical Analysis 1: Comparison: Me & My Wishes Intervention/Group 1 vs Me & My Wishes Wait-list Control/Group 2; Test type: Superiority; p = .081, Mixed Models Analysis; Mean Difference (Final Values) = .09, 95% CI 2-sided [-.01 to .19]

6. Other Pre Specified Outcome: Concordance of End of Life Preferences, Video and Family
Description: EOL preferences include treatment preferences (cardiopulmonary resuscitation, or CPR; breathing machine; tube feeding; life support; and pain treatment). Preferences from the videos and surveys were coded as yes, no, don't know, or missing. Concordance occurred when the coded preferences in the resident's video and family member response matched.
Time Frame: Baseline, time of sharing (within 3 months of baseline), and 90 days post sharing video
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Me & My Wishes Intervention/Group 1 | Me & My Wishes Wait-list Control/Group 2
Number analyzed (Participants) | 17 | 19
percentage of agreement
  Baseline | 48.15 (23.04) | 38.26 (35.63)
  Time of Sharing | 60.80 (23.44) | 62.61 (26.49)
  90 days | 53.91 (17.51) | 52.63 (24.23)
Statistical Analysis 1: Comparison: Me & My Wishes Intervention/Group 1 vs Me & My Wishes Wait-list Control/Group 2; Test type: Superiority; p = .033, Mixed Models Analysis; Mean Difference (Final Values) = .21, 95% CI 2-sided [.11 to .3] — Calculation of mean differences were derived from mixed model analyses

ADVERSE EVENTS:
Time Frame: baseline to end of study (6-9 months)
Groups:
- Me & My Wishes Intervention/Group 1 Family: In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline with family.
- Me & My Wishes Wait-list Family: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be produced and viewed within three months with family.
- Me & My Wishes Intervention Group 1 Staff: In Group 1 (early intervention group) NHs, video recording, editing, and viewing will occur within three months of baseline with staff
- Me & My Wishes Control/Group 2 Staff: In Group 2 (delayed sharing) NHs, residents will be on a wait-list; after the delayed start, their video will be produced and viewed within three months with staff
Arm/Group | Me & My Wishes Intervention/Group 1 Resident | Me & My Wishes Wait-list Control/Group 2 Resident | Me & My Wishes Intervention/Group 1 Family | Me & My Wishes Wait-list Family | Me & My Wishes Intervention Group 1 Staff | Me & My Wishes Control/Group 2 Staff
All-Cause Mortality (participants affected / at risk) | 2/26 | 1/24 | 0/25 | 0/25 | 0/13 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/25 | 0/25 | 0/13 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/25 | 0/25 | 0/13 | 0/25

LIMITATIONS AND CAVEATS:
Randomization at site level and despite, randomizing in blocks, our sites differed. Small sample size: Primary outcome (goals of care conversations) without the power to detect statistical significance. Findings may be muted or underestimated because we measured documentation; conversations may occur without being documented. Majority of participants being of one racial group (white) and one geographic region limits generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03861429/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03861429/SAP_002.pdf
  • Informed Consent Form (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03861429/ICF_000.pdf